CLINICAL TRIAL: NCT05030701
Title: Toxicity of Treatments for Non-tuberculous Mycobacterial Infections in Cancer Patients or Not
Acronym: MYCATRES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0072
Record Dates: First submitted 2021-07-13; First posted 2021-09-01 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Mycobacterium; Cancer; Treatment Side Effects
Keywords: Mycobacterium; cancer; Treatment Side Effects
MeSH Terms: conditions — Mycobacterium Infections; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cancerous patients
- non cancerous patients

SUMMARY:
Non-tuberculous mycobacteria (NTM) are increasingly common and have a poor prognosis: 5-year mortality can reach 40 to 50%, depending on the type of mycobacteria and the immune system of the host involved. Cancer patients are at higher risk of infectious morbidity and mortality, which may be due to disease-related immune dysfunction, immunosuppressive effects of chemotherapy, or long-term placement of a vascular catheter. However, data on the treatment of NTM species that cause infections and the disease characteristics of these pathogens in cancer patients are limited despite the growing cancer population worldwide. Recently, M. avium infections have been described in patients suffering from cancers (hematological or not), in particular in patients receiving checkpoint inhibitors. Although the proportion of M. avium pneumonia in retrospective series is low (0.8-2%), it has been shown that this population is younger, suffers less from sub-pulmonary pathology. (indicating immunosuppression in these patients) but are therefore treated less than non-cancerous subjects.

This retrospective study in CHU Amiens is searching on the number of side effects of NTM treatment in two groups (cancerous and no cancerous) to assess the cause of the decrease of NTM treatment in cancerous patients.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or more than 18 years18
* Patients diagnosed by an infection with non-tuberculous mycobacteria according to ATS guidelines.
* Patients received the NTM treatment.

Exclusion Criteria:

* age less than 18 years
* Patients diagnosed by NTM without treatment.
* Patients with a positive sample of NTM but without infection.
* Exclusion of other disorders such as tuberculous.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients infected with Nontuberculous mycobacteria, collected from CHU Amiens 2015 to 2020, extracted from the medical information service by the RUM (medical unit summary) with a diagnostic code ICD-10 which is the International Classification of diseases, commonly known as the international statistical classification of diseases and related health problems and Chapters A31.0, A31.8, A31.9.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
variation of side effects number of non-tuberculous mycobacteria treatment between cancerous and non cancerous patient groups. | 3 months
  The main objective of this study is to determine the number of side effects of the treatment of non-tuberculous mycobacteria in patients with this infection with or without cancer at the CHU Picardie Amiens.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No